CLINICAL TRIAL: NCT02851095
Title: A Single-Dose, Open-Label, Randomized, 4-Way Crossover Pivotal Study to Assess the Bioequivalence of the Metformin Component of the Fixed Dose Combination Tablet of Canagliflozin and Metformin Extended Release (XR) 1 x (50 mg/1000 mg) With Respect to the Metformin XR Tablet (Locally Sourced From Canada [GLUMETZA, 2 x 500 mg]) Coadministered With Canagliflozin (1 x 50 mg) in Healthy Fed and Fasted Subjects
Brief Title: A Study to Assess the Bioequivalence of the Metformin Component of the Fixed Dose Combination Tablet of Canagliflozin and Metformin Extended Release (XR) With Respect to Metformin XR Tablet Coadministered With Canagliflozin in Healthy Fed and Fasted Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108199; 28431754DIA1074 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence ADBC (Experimental): Participants will receive Treatment A (1 canagliflozin tablet 50 milligram (mg) along with two Extended Release (XR) tablet of metformin of each 500 mg orally under fed condition) on Day 1 of treatment period 1, then Treatment D of (1 XR fixed dose combination [FDC] tablet containing canagliflozin 50 mg and metformin 1000 mg orally under fasted condition) on Day 1 of treatment period 2, then Treatment B (1 XR FDC tablet containing canagliflozin 50 mg and 1 metformin 1000 mg orally under fed condition) on Day 1 of treatment period 3, followed by Treatment C (1 canagliflozin tablet 50 mg along with 2 metformin (XR) tablets of each 500 mg orally under fasted condition) on Day 1 of treatment period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin and Metformin Extended Release (XR) Fixed Dose Combination [FDC]; Drug: Canagliflozin; Drug: Metformin Extended Release (XR)
- Treatment Sequence BACD (Experimental): Participants will receive Treatment B on Day 1 of treatment period 1, then Treatment A on Day 1 of treatment period 2, then Treatment C on Day 1 of treatment period 3, followed by Treatment D on Day 1 of treatment period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin and Metformin Extended Release (XR) Fixed Dose Combination [FDC]; Drug: Canagliflozin; Drug: Metformin Extended Release (XR)
- Treatment Sequence CBDA (Experimental): Participants will receive Treatment C Day 1 of treatment period 1, then Treatment B on Day 1 of treatment period 2, then Treatment D on Day 1 of treatment period 3, followed by Treatment A on Day 1 of treatment period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin and Metformin Extended Release (XR) Fixed Dose Combination [FDC]; Drug: Canagliflozin; Drug: Metformin Extended Release (XR)
- Treatment Sequence DCAB (Experimental): Participants will receive Treatment D on Day 1 of treatment period 1, then Treatment C on Day 1 of treatment period 2, then Treatment A on Day 1 of treatment period 3, followed by Treatment B on Day 1 of treatment period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin and Metformin Extended Release (XR) Fixed Dose Combination [FDC]; Drug: Canagliflozin; Drug: Metformin Extended Release (XR)

INTERVENTIONS:
Drug: Canagliflozin and Metformin Extended Release (XR) Fixed Dose Combination [FDC] — Participants will receive 1 XR FDC tablet containing canagliflozin 50 mg and metformin 1000 mg orally under fed (Treatment B) or fasted (Treatment D) condition in a given treatment period as per treatment sequence.
Drug: Canagliflozin — Participants will receive canagliflozin 50 mg oral tablet) under fed (part of treatment A) or fasted (part of treatment C) condition in a given treatment period as per treatment sequence.
Drug: Metformin Extended Release (XR) — Participants will receive 2 metformin XR tablets of each 500 mg orally under fed (part of treatment A) or fasted (part of treatment C) condition in a given treatment period as per treatment sequence.

SUMMARY:
The purpose of this study is to evaluate bioequivalence of the metformin component of the Fixed Dose Combination (FDC) tablet compared with the metformin Extended Release (XR) tablets co-administered with canagliflozin in healthy fed and fasted participants.

ELIGIBILITY:
Inclusion Criteria:

* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies
* Before randomization, a woman must be either Not of childbearing potential or of childbearing potential and agrees to use a highly effective method of contraception (failure rate of less than [<]1 percent [%] per year when used consistently and correctly) throughout the study
* All women must have a negative urine pregnancy test at Screening and on Day -1 of each Treatment Period
* Body mass index (BMI) (weight [kg]/height^2 [m]2) between 18 and 30 kg/m^2 (inclusive), and body weight not less than 50 kilogram (kg)
* Blood pressure between 90 and 140 millimeter of mercury (mmHg), inclusive, systolic and no higher than 90 mmHg diastolic at Screening or Day -1 of each Treatment Period
* Normal renal function evidenced by estimated Glomerular Filtration Rate (eGFR) greater than or equal to (>=90) milliliters per minute (mL/min)/1.73m^2 using the Modification of Diet in Renal Disease Study (MDRD) equation as defined in the protocol

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis as assessed by the investigator at Screening or Day -1 of the first Treatment Period
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) (Screening only) as assessed by the investigator at Screening or on Day -1 of the first Treatment Period as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, hormonal contraceptives and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled
* History of, or a reason to believe a participant has a history of drug or alcohol abuse within the past 5 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Metformin | Pre-dose, 0.5 hour (hr), 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, hr post dose on Day 1; 24 hr post-dose on Day 2
  The Cmax is the maximum observed plasma concentration of metformin.
Area Under the Plasma Concentration Time Curve From Time 0 to The Time of the Last Observed Quantifiable Concentration (AUClast) of Metformin | Pre-dose, 0.5 hour (hr), 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, hr post dose on Day 1; 24 hr post-dose on Day 2
  The AUClast is the area under the plasma concentration time curve from time 0 to the time of the last observed quantifiable concentration (Clast).
Area Under the Plasma Concentration Time Curve From Time 0 to Infinite Time [AUC (0-infinity)] of Metformin | Pre-dose, 0.5 hour (hr), 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, hr post dose on Day 1; 24 hr post-dose on Day 2
  The AUC (0-infinity) is the area under the plasma concentration time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Day -1 to End of study (up to 58 Days)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Lincoln, Nebraska, United States